CLINICAL TRIAL: NCT01600248
Title: Online Chronic Pain Therapy for Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H2012:078
Record Dates: First submitted 2012-05-10; First posted 2012-05-17 (Estimated); Last update posted 2015-08-21 (Estimated); Status verified 2015-08

CONDITIONS: Chronic Pain
Keywords: Chronic Pain; Military; Veteran; Online; Acceptance
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment arm (Other): This is an open-label pilot study with no control group. Participants pre-treatment scores are compared to their post-treatment scores.
  Interventions: Behavioral: Online ABBT for Chronic Pain in Military

INTERVENTIONS:
Behavioral: Online ABBT for Chronic Pain in Military — Participants will complete an 8-module, self-paced, online program for chronic pain using Acceptance-Based Behavioural Therapy (ABBT) as the therapeutic modality.

SUMMARY:
This study will evaluate the usefulness of an online, self-directed treatment for chronic pain that has been designed specifically for individuals who are currently or have previously served in the military.

DETAILED DESCRIPTION:
This study will evaluate the efficacy of an eight-module, online, self-directed treatment for chronic pain using Acceptance-Based Behavioural Therapy (ABBT) as the treatment modality. The online modules are tailored to the unique issues of individuals with a military background. The modules will be delivered via the WebCAPSI Therapy program, an online, password-protected program that allows participants to anonymously progress through all modules at their own pace. ABBT modules cover the following: Introduction, Acceptance, Values, Cognitive Defusion, Mindfulness, Exercise/Pacing/Communication Skills, Self-as-Context, and Willingness. Modules encourage understanding of the information through audio files, military-specific vignettes, written materials, and homework exercises. Modules are designed to be completed in 60 minutes or less. Participants will have access to the online treatment for a three month period and will be encouraged to complete one module per week.

ELIGIBILITY:
Inclusion Criteria:

* Chronic pain condition of duration 6 months or longer
* Patient at OSI Clinic in Winnipeg
* Access to a computer with internet at least once per week for 60 minutes

Exclusion Criteria:

* Active psychosis
* Actively suicidal
* Unstable living conditions
* Seriously impaired concentration
* Inability to read and write in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2012-06; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline in McGill Pain Questionnaire - Short Form | 8 weeks
  A brief self-report questionnaire that measures sensory and affective components of clinical pain.
Change from baseline in Chronic Pain Acceptance Questionnaire - Revised | 8 weeks
  A 20-item measure of acceptance of chronic pain with items scored from "0 = Never true" to "6 = Always true".
Change from baseline in Pain Catastrophizing Scale | 8 weeks
  One of the most widely used instruments for measuring catastrophic thinking related to pain. A 13-item measure with items rated from "0 = Not at all" to "4 = All the time."
Change from baseline in Tampa Scale for Kinesiophobia | 8 weeks
  A self-report measure of fear of movement and/or re-injury. 17 items rated from "1 = strongly disagree" to "4 = strongly agree"
Change from baseline in Pittsburgh Sleep Quality Index | 8 weeks
  A self-rated questionnaire which assesses sleep quality and disturbances over a 1-month time interval

SECONDARY OUTCOMES:
Client Satisfaction Questionnaire | At completion of module, approximately 8 weeks
  An eight item questionnaire regarding client satisfaction with the treatment.
Change from baseline in Beck Depression Inventory - Second Edition | 3 months
  A 21 item self-report measure of severity of depressive symptoms.
Change from baseline in Beck Anxiety Inventory | 3 months
  A 21-item self-report measure assessing severity of symptoms of anxiety
Change from baseline in PTSD Checklist - Military Version | 3 months
  A 17-item self-report measure assessing severity of PTSD symptoms related to stressful military experiences.

CONTACTS AND LOCATIONS:
Overall Officials: Pamela L Holens, Ph.D., Principal Investigator — University of Manitoba
Locations (1):
- OSI Clinic, Deer Lodge Centre, Winnipeg, Manitoba, Canada